CLINICAL TRIAL: NCT00497042
Title: Safety and Efficacy of Using the Endodontic Self Adjusting File - SAF for Root Canal Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ReDent Nova (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-07-AS-030-CTIL
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2007-07-11 (Estimated); Status verified 2007-07

CONDITIONS: Teeth, Endodontically-Treated
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Self Adjusting File

SUMMARY:
The study's primary goal is to assess the safety of the SAF (Self Adjusting File) device for root canal treatments.

The study's secondary goal is to evaluate the effectiveness of the SAF device for root canal treatments

DETAILED DESCRIPTION:
Endodontic treatment (root canal treatment) is conducted when the dental pulp is inflamed or when it becomes necrotic and infected. The main cause for both these cases is dental caries and they represent sequential stages of the same disease with inflammation preceding the necrosis and infection.

Mechanically, both conditions are treated in a rather similar manner, by "cleaning and shaping", using endodontic files and irrigation solutions. This mechanical process is aimed to thoroughly disinfect the root canal by removing all tissue remnants while enlarging the diameter of the root canal, to remove all canal irregularities that may harbor bacteria. During this process an inner layer of dentin has to be removed from all the surface of the root canal. A second goal of root canal treatment is to allow adequate sealing of the canal space by a root canal filling, in order to prevent future bacterial contamination. For teeth with inflamed vital pulps, once this stage is completed the root canal may be sealed. When necrotic infected root canals are involved, this stage greatly reduces the bacterial load in the canal but an additional stage of disinfection by medicaments, sealed in the canal until the next appointment, may be required.

The SAF file is an endodontic file designed to be operated by a Profin dental low-speed hand-piece (W&H, Burmoos / Salzburg, Austria), which converts rotation into a transline reciprocal movement. The active part of the file is manufactured from a thin-walled tube of medical grade nickel-titanium alloy. It has a cylindrical shape and can be compressed to allow its insertion into thin root canal, due to its lattice-like structure.

The SAF file is an endodontic file of a revolutionary design. As any endodontic file it is designed to remove dentin from the root canal walls and enlarge the canal. Its advantages are:

* it grinds the inner root canal wall, rather than machine-cut it,
* it adapts itself to the cross section of the canal and enlarges it to a wider version of its original form.
* It enlarges the canal; using one instrument which gradually expands in size, rather than tediously using a sequence of instruments.
* Its hollow space allows for continuous irrigation and flushing out the ground material rather than tediously stopping again and again to remove the instrument from the root canal and flush it, and
* it is highly resistant to breakage

The tested device is an engine-operated endodontic file used for root canal treatment. It is constructed from a medical grade nickel-titanium alloy and designed as a hollow tube made of a delicate metal lattice, attached to a dental hand-piece. It is operated in root canals with a continuous rinsing. The rinsing solution enters the hollow device through a special irrigator attachment, flows through the root canal and emerges through the access cavity, where it is collected using a dental suction tip.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects is 18 years or older
2. Subject has one or more teeth that have to go through a root canal treatment
3. Roots are fully formed and with a mature apex
4. At least one of the roots to be treated has periapical radiolucency with a diameter of 2-6mm and a PAI score of 4 or 5
5. Subject had signed the informed consent form

Exclusion Criteria:

1. Previous root canal filling
2. Roots with abnormal root canal anatomy
3. Roots for which a good quality periapical radiographic image cannot be produced
4. Un-restorable teeth
5. Significant periodontal pockets
6. Patients who are pregnant or breast-feeding
7. Uncontrolled systemic hypertension
8. Severe uncontrolled Diabetes Mellitus
9. Current steroid therapy in excess of prednisone 5 mg/day
10. HIV positive patients
11. Hepatitis
12. Chronic renal failure
13. Hematological disease (malignancy, severe anemia)
14. Osteoporosis, receiving biphosphonates
15. Post head and neck irradiation treatment
16. Other severe or life-threatening systemic disease
17. Known cognitive disorder, psychiatric and/or neurological disease
18. Concurrent participation in any other clinical study
19. Patients cannot understand or not willing to sign the informed consent
20. During chemotherapy or radiology treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)

PRIMARY OUTCOMES:
Treatment related operative and postoperative major complications. | One year.

SECONDARY OUTCOMES:
Healing of pariapical leasions as a result of the endodontic treatment. | One year.

CONTACTS AND LOCATIONS:
Overall Officials: Amnon Singer, DMD, Principal Investigator — Redent Nova Ltd.
Locations (1):
- Tel Aviv Souraski Medical Center, Tel Aviv, Israel